CLINICAL TRIAL: NCT04357119
Title: Evaluation on Common Limb Length in Laparoscopic One-anastomosis Gastric Bypass for Morbidly Obese Patients
Brief Title: Common Limb Length in One-anastomosis Gastric Bypass
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hosam Hamed, Lecturer of general surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MD/16.05.65
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Obesity, Morbid; Weight Loss; Bariatric Surgery Candidate
Keywords: One-anastomosis gastric bypass; Common limb length; Bariatric surgery; Malnutrition
MeSH Terms: conditions — Obesity, Morbid; Weight Loss; Malnutrition

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CL measured from Treitz ligament (Active Comparator): A 14-16 cm long gastric tube is created using a 60 mm stapler starting on the lesser curvature at the crow's foot level. It is tailored following the edge of a 38F calibrating orogastric tube up to the angle of His. A loop gastroenterostomy is then created with the small bowel about 200 cm distal to the ligament of Treitz with the same stapler using a 60 mm blue cartridge
  Interventions: Procedure: One-anastomosis gastric bypass
- CL measured from ileocecal valve (Active Comparator): A 14-16 cm long gastric tube is created using a 60 mm stapler starting on the lesser curvature at the crow's foot level. It is tailored following the edge of a 38F calibrating orogastric tube up to the angle of His. A loop gastroenterostomy is then created with the small bowel about 300 cm proximal to the ileocecal valve with the same stapler using a 60 mm blue cartridge
  Interventions: Procedure: One-anastomosis gastric bypass

INTERVENTIONS:
Procedure: One-anastomosis gastric bypass — Laparoscopic single anastomosis gastric bypass is reported to be a safe alternative to LRYGB, showing comparable efficacy in weight reduction and resolution of metabolic complications with reduced surgical complications.
  The advantages with this technique as claimed by those speaking in favor of it are many: fewer sites for leakage and internal hernia, easier and faster to learn and perform, easy to reverse and revise, and with results at least comparable with the result following standard Roux-en-Y gastric bypass (RYGB).
  The length of the biliopancreatic limb in single anastomosis gastric bypass as reported by Rutledge is fixed 200 cm starting at the duodenojejunal junction, neglecting the length of the common limb.
  Because of deficient data regarding the effect of common limb length on the outcome of LSAGB, so a clinical trial shall add new knowledge regarding sufficient weight loss, rate of complications and the need for revision.

SUMMARY:
Evaluation of the effect of the common limb length on the outcome of laparoscopic single anastomosis gastric bypass in morbidly obese patients.

Two groups of patients: one group with a common limb length of about 200 cm distal to the ligament of Treitz and the second group with a common limb length of 300 cm proximal to the ileocecal valve.

Groups are evaluated regarding percentage of excess weight loss, resolution of comorbidities, and long term complications.

DETAILED DESCRIPTION:
The present study is a prospective, randomized comparative clinical trial involving 60 patients (due to limited flow rate and high expenses [14]) who will be subjected to laparoscopic single anastomosis gastric bypass at the department of surgery, Mansoura university, Mansoura, Egypt at the period from May 2016 to May 2019.

Patients will be randomly allocated into 2 groups with 30 patients undergoing LSAGB with measuring two meters from the duodenojejunal junction, and the other 30 undergoing LSAGB with measuring three meters from the ileocecal valve.

Informed consent will be obtained from all patients participating in the study after explaining the patients about the benefits and the potential risks involved.

Inclusion criteria:

1. Morbid obesity with BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 associated with one or more co-morbidities (type 2 diabetes, arterial hypertension, sleep apnea, dyslipidemia, arthritis).
2. Age between 18 and 60 years old.

Exclusion criteria:

1. Pregnancy or desire to be pregnant during the study.
2. Abnormal findings on upper GI endoscopy.
3. Presence of chronic diarrhea (≥ 3 liquid or loose stools per day, over a period of more than 4 weeks).
4. Obesity due to organic disease e.g, cushing disease and hypothyroidism.
5. Previous bariatric surgery.
6. Coexisting severe hepatic, pulmonary, renal, cardiovascular, neurological and psychiatric diseases.

Subjects and preoperative evaluation:

Preoperative evaluation including

* Clinical history.
* Thorough Physical examination.
* BMI is calculated as weight in kilogram divided by height in metre2.
* Routine laboratory tests and urinalysis. Throid function and serum cortisol done to rule out organic illness.
* Fasting blood sugar, HbA1c and lipid profile.
* ABG and pulmonary function routinely done for all patients preoperative.
* Fecal fat excretions done to follow up incidence of steatorrhea.
* Imaging studies (chest radiograph and ultrasound abdomen).
* Routine upper GI endoscopy will be done preoperative.

Outcomes:

The primary outcome measures excess weight loss % one and 2 years after surgery.

Secondary outcomes measures:

* Weight loss according to the absolute weight loss (time frame: 1, 3, 6, 12, 18 and 24 months after surgery).
* Waist size reduction according to the absolute waist size (time frame: 1, 3, 6, 12, 18 and 24 months after surgery).
* Medical and surgical complication (anastomotic leaks, biliary reflux, bowel obstruction, anastomotic ulcers, anastomotic stenosis, chronic gastritis, esophagitis, iron deficiency anemia) followed at 1, 12 and 24 months after surgery.

Early complications are detected during the 1st month following surgery while late complications defined from 1 to 24 months after surgery.

* Improvement in glycemic parameters (HbA1C, Fasting blood sugar, Post lunch blood sugar).
* Remission of hypertension and lipid profile changes.
* Patient's quality of life 6, 12, 24 months after surgery (according to the Bariatric Analysis and Reporting Outcome System questionnaire "BAROS").
* Frequency of diarrhea based on the gastrointestinal quality of life index (GIQLI) questionnaire.
* Rate of revision due to intolerable complications, or due to insufficient weight loss.

The outcomes will be planned to be monitored and analyzed at 3 months interval for 24 months.

Prevention of surgical site infection and perioperative antiplatelet drug administration will be managed according to validated criteria [15, 16].

Surgical technique:

Patients are placed in the reverse Trendelenburg position with legs spread. The surgeon stands between patient's legs. The monitor is at the head of the operating-table to the left side of the patient. We always use a 30_ optic and five trocars.

The technique used for LSAGB has been described [16]. A 14-16 cm long gastric tube is created using a 60 mm stapler starting on the lesser curvature at the crow's foot level. It is tailored following the edge of a 38F calibrating orogastric tube up to the angle of His. A loop gastroenterostomy is then created with the small bowel about 200 cm distal to the ligament of Treitz with the same stapler using a 60 mm blue cartridge for the first group and about 300cm proximal to the ileocecal valve for the second group. The gastrojejunal anastomosis is then closed with a double-layer locking running 2-0 suture. All patients are checked by an intraoperative methylene blue test at the end of the procedure. A drain tube is placed in all the patients.

Postoperative care:

All the patients are monitored in the recovery room and transferred to the wards or to the intensive care unit when needed. Early postoperative ambulation is strongly encouraged with patients getting out of bed the evening of the surgery and walking by postoperative day 1. A clear liquid diet started on day 2, and advanced to pureed food 1 week later, and to solid food by the fourth postoperative week. At discharge the drain is removed and detailed dietary instructions provided to the patients. Patients are advised to take daily multivitamins and supplemental minerals, as well as proton pomp inhibitor (PPI) prophylaxis for 6 months. Follow-up scheduled at 1, 3, 6, 12, and 24 months postoperatively, then twice a year.

Statistical analysis will be performed using the SPSS 19 system (SPSS Inc., Chicago, IL, United States). Continuous data will be expressed as the mean ± SD, and categorical variables expressed as the percent changes. Statistical significance defined as P values < 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. Morbid obesity with BMI ≥ 40 kg/m2 or BMI ≥ 35 kg/m2 associated with one or more co-morbidities (type 2 diabetes, arterial hypertension, sleep apnea, dyslipidemia, arthritis).
2. Age between 18 and 60 years old.

Exclusion Criteria:

1. Pregnancy or desire to be pregnant during the study.
2. Abnormal findings on upper GI endoscopy.
3. Presence of chronic diarrhea (≥ 3 liquid or loose stools per day, over a period of more than 4 weeks).
4. Obesity due to organic disease e.g, cushing disease and hypothyroidism.
5. Previous bariatric surgery.
6. Coexisting severe hepatic, pulmonary, renal, cardiovascular, neurological and psychiatric diseases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
the percentage of excess weight loss | 2 years
the percentage of total body weight loss | 2 years
resolution or improvement of comorbidities | 2 years
  cessation of treatment or reduction of medications

SECONDARY OUTCOMES:
early postoperative morbidities | 3 months
  leakage, bleeding, thromboembolic complications
late complications | 2 years
  malnutrition, hernia, anastomotic ulcer

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Shoma, Study Director — Head of Unit 7 , Department of Surgery

IPD SHARING:
Plan to Share IPD: Yes
The data are planned to be published as a research paper.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: The data is panned to be published as a research paper in one of the journals concerned with obesity surgery
Access Criteria: The data is planned to be available on the journal that the research paper will be submitted to